CLINICAL TRIAL: NCT03201068
Title: Impact of a Probiotic Supplement on the Microbiome, Immune System, and Metabolic Syndrome
Brief Title: Probiotic Supplement and Microbiome, Immune System and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Clorox Company (Unknown)
Responsible Party: Principal Investigator, Justin L. Sonnenburg, Associate Professor of Microbiology and Immunology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 41697
Record Dates: First submitted 2017-06-23; First posted 2017-06-28 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Syndrome; Microbiome; Immune Function; Inflammation
MeSH Terms: conditions — Metabolic Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic supplement (Experimental): Renew Life Formulas, Inc
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — Probiotic supplement capsule
  Other Names: Renew Life Formulas, Inc
  Arms: Probiotic supplement
Dietary Supplement: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
This study will define the impact of a probiotic supplement on microbiome, immune system, and metabolic syndrome. This study will determine the degree to which a probiotic supplement can 1) improve metabolic markers and metrics of metabolic syndrome, 2) alter microbiota composition and function, 3) impact microbiota metabolites, short-chain fatty acids-potential normalizers of metabolic and immune dysfunction, and 4) regulate immune status and function including reducing chronic, systemic inflammation as assessed by high dimensional immune profiling.

DETAILED DESCRIPTION:
The centrality of the gut microbiota to human health has emerged in just the last decade, with the last three years implicating our modern, deteriorated gut microbiota in numerous chronic diseases. It is likely dietary changes in the last half-century consistent with adoption of the Western diet have had an adverse impact on the gut microbiota. A critically important next step in this field of research is to identify how different probiotic supplements can potentially restore the microbiota in alignment with the optimization of human health, particularly in regard to the reversal or prevention of chronic diseases including obesity, metabolic syndrome, and inflammatory bowel disease. This study is designed to elicit and contrast the amount of increase in microbiota diversity and related metabolic output achievable following consumption of a probiotic supplement commonly available to the general population. The results could contribute to dietary recommendations for reversing the chronic disease epidemics of westernization.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older
* Must have metabolic syndrome as defined by having at least 2 of the 5 criteria per either ATP III guidelines OR International Diabetes Federation (IDF) guidelines:

ATP III guidelines:

1. Abdominal obesity, defined as a waist circumference in men ≥102 cm (40 in) and in women ≥88 cm (35 in)
2. Serum triglycerides ≥150 mg/dL (1.7 mmol/L) or drug treatment for elevated triglycerides
3. Serum high-density lipoprotein (HDL) cholesterol <40 mg/dL (1 mmol/L) in men and <50 mg/dL (1.3 mmol/L) in women or drug treatment for low HDL cholesterol
4. Blood pressure ≥130/85 mmHg or drug treatment for elevated blood pressure
5. Fasting plasma glucose (FPG) ≥100 mg/dL (5.6 mmol/L) or drug treatment for elevated blood glucose

International Diabetes Federation Guidelines:

1. Increased waist circumference, with ethnic-specific waist circumference cut-points:

   White and all other ethnic groups - Men ≥ 94 cm; Women ≥ 80 cm South Asians, Chinese, and Japanese - Men ≥ 90 cm; Women ≥ 80 cm

   PLUS any two of the following:
2. Triglycerides ≥150 mg/dL (1.7 mmol/L) or treatment for elevated triglycerides
3. HDL cholesterol <40 mg/dL (1.03 mmol/L) in men or <50 mg/dL (1.29 mmol/L) in women, or treatment for low HDL
4. Systolic blood pressure ≥130, diastolic blood pressure ≥85, or treatment for hypertension
5. FPG ≥100 mg/dL (5.6 mmol/L) or previously diagnosed type 2 diabetes; an oral glucose tolerance test is recommended for patients with an elevated fasting plasma glucose, but not required.

Exclusion Criteria:

* Body Mass Index (BMI) ≥ 40
* LDL >160 mg/dL.
* Vital signs outside of acceptable range at Screening Visit: blood pressure >159/99, oral temperature ≥ 100°F, pulse >100.
* Use of any of the following drugs within the last 6 months:systemic antibiotics (must be discontinued and avoided for 2 months prior to the study start), antifungals, antivirals or antiparasitics (intravenous, intramuscular, or oral); oral, intravenous, intramuscular, nasal or inhaled corticosteroids; cytokines; methotrexate or immunosuppressive cytotoxic agents;
* Use of large doses of commercial probiotics consumed within the last 6 months (greater than or equal to 108 cfu or organisms per day) - includes tablets, capsules, lozenges, chewing gum or powders in which probiotic is a primary component (must be discontinued and avoided for one month prior to the study start). Ordinary dietary components such as fermented beverages/milks, yogurts, foods do not apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Metabolic syndrome parameters: Waist Circumference, Blood pressure, Triglycerides, HDL-cholesterol, and Fasting Glucose. | Baseline (week 4) and end of intervention (week 14)
  10-week change from Baseline (week 4) in the number of subjects presenting 3 of the 5 parameters for metabolic syndrome (waist circumference, blood pressure, triglycerides, HDL-cholesterol, and fasting glucose) at 14 weeks (end of intervention).

SECONDARY OUTCOMES:
Microbiota composition | Baseline (week 4) and end of intervention (week 14)
  10-week change from baseline (week 4) in 16S rRNA enumeration at 14 weeks (end of intervention), determined using Illumina-based sequencing.
Microbiota metabolites | Baseline (week 4) and end of intervention (week 14)
  10-week change from Baseline (week 4) in short-chain fatty acids (SCFA) at 14 weeks (end of intervention).
Cytokines | Baseline (week 4) and end of intervention (week 14)
  10-week change from Baseline (week 4) in cytokines at 14 weeks (end of intervention).
Chemokines | Baseline (week 4) and end of intervention (week 14)
  10-week change from Baseline (week 4) in chemokines at 14 weeks (end of intervention).
hs-C Reactive Protein (CRP) | Baseline (week 4) and end of intervention (week 14)
  10-week change from Baseline (week 4) in hs-CRP at 14 weeks (end of intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wastyk HC, Perelman D, Topf M, Fragiadakis GK, Robinson JL, Sonnenburg JL, Gardner CD, Sonnenburg ED. Randomized controlled trial demonstrates response to a probiotic intervention for metabolic syndrome that may correspond to diet. Gut Microbes. 2023 Jan-Dec;15(1):2178794. doi: 10.1080/19490976.2023.2178794. PMID 36803658
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/ProjectProbiotic.html